CLINICAL TRIAL: NCT04466111
Title: A Post-Market, Observational Clinical Study to Evaluate the Effects of Differential Target Multiplexed DTM™ SCS Programming in Treating Intractable Chronic Upper Extremity Limb Pain
Brief Title: Observational, Post Market Study in Treating Chronic Upper Extremity Limb Pain
Acronym: PROC2020PM
Status: Completed | Type: Observational
Sponsor: SGX Procura LLC (Industry)
Responsible Party: Sponsor
Organization: SGX Medical LLC (Industry)
Other Study IDs: DTM-PROC-2020PM3
Record Dates: First submitted 2020-07-06; First posted 2020-07-10 (Actual); Results first posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-03

CONDITIONS: Upper Limb; Pain
Keywords: upper limb; Spinal Cord Stimulation; Pain
MeSH Terms: conditions — Pain | interventions — Spinal Cord Stimulation; Drug Delivery Systems

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Intellis neurostimulator system — The study will use the commercially available IntellisTM neurostimulator and compatible SCS system components from Medtronic using stimulation parameters within the specifications approved for use in the approved indications. The study will stimulate the cervical dorsal columns of the spinal cord.
  Other Names: Spinal Cord Stimulation (SCS) device system

SUMMARY:
This is a post-market, open-label, prospective, multi-center, observational study evaluating upper limb pain relief with the DTM™ SCS programming approach.

Data at follow-up visits will be compared to baseline assessments collected at the beginning of the study.

DETAILED DESCRIPTION:
This is a post-market, open-label, prospective, multi-center, observational study evaluating upper limb pain relief with the DTM™ SCS programming approach.

Data at follow-up visits will be compared to baseline assessments collected at the beginning of the study.

The expected total duration of this study is approximately 26 months. Enrollment of participants is expected to last 20 months. Participants that have received the permanent implant will be followed up for 12 months after their device has been activated. A participant will likely be committed to the study for about 14 months. This consists of Baseline assessments, up to 10 days of trial stimulation, and 12 months of treatment following implantation and activation of the device. All subjects who plan on remaining implanted through the 6-month visit or who have completed their 6-month visit will be offered to return for an additional 12-month visit. This would increase their commitment to the study to 14 months.

ELIGIBILITY:
Inclusion Criteria:

* A subject must MEET ALL of the following inclusion criteria:

  1. Be diagnosed with chronic, intractable pain of the upper limb related to the cervical spine and/or neuropathic arm pain.
  2. Be a candidate for SCS system (trial and implant) per labeled indication (upper limb pain due to one of the conditions listed in indications statement)
  3. Considering daily activity and rest, has average upper limb pain intensity of ≥ 5 out of 10 cm on the Visual Analog Scale (VAS) at enrollment
  4. Be willing and capable of giving written informed consent to participate in this clinical study based on voluntary agreement after a thorough explanation of the subject's participation has been provided.
  5. Be willing and capable of subjective evaluation, read and understand written questionnaires, and read, understand and sign the written inform consent.
  6. Be 18 years of age or older at the time of enrollment
  7. Be on a stable pain medication regime, as determined by the study investigator, for at least 30 days prior to enrolling in this study
  8. Be willing and able to comply with study -related requirements, procedures, and visits, including not increasing pain meds through the three month visit
  9. Has adequate cognitive ability to use a patient programmer and recharger as determined by the Investigator

Exclusion Criteria:

* A subject must NOT MEET ANY of the following exclusion criteria:

  1. Has a medical, anatomical, and/or psychosocial condition that is contraindicated for commercially available IntellisTM SCS systems as determined by the Investigator
  2. Have a medical condition or pain in other area(s), not intended to be treated with SCS, that could interfere with study procedures, as determined by the Investigator
  3. Currently enrolled or planning to enroll in an interventional clinical study that could potentially confound the study results (co-enrollment in an interventional study is only allowed when documented pre-approval is obtained from the study manager or designee)
  4. Has an existing active implanted device such as a pacemaker, another SCS unit, peripheral nerve stimulator, and/or drug delivery pump.
  5. Has pain in other area(s) and/or medical condition requiring the regular use of significant pain medications that could interfere with accurate pain reporting, study procedures, and/or confound evaluation of study endpoints, as determined by the Investigator
  6. Has significant cervical stenosis, as determined by the Investigator
  7. Has facet spondylosis, as determined by the Investigator
  8. Has mechanical spine instability, as determined by the Investigator
  9. Has undergone, within 30 days prior to enrollment, an interventional procedure and/or surgery to treat upper limb pain, which is providing significant pain relief
  10. Has unresolved major issues of secondary gain (e.g., social, financial, legal, such as worker compensation matters)
  11. Be pregnant as determined by urine testing unless female subject is surgically sterile or post-menopausal. If female, sexually active, and childbearing age, subject must be willing to use a reliable form of birth control.
  12. Have evidence of an active disruptive psychological or psychiatric disorder as determined by a psychologist
  13. Have a current diagnosis of a progressive neurological disease as determined by the Investigator
  14. Have a current diagnosis of a coagulation disorder, bleeding diathesis, progressive peripheral vascular disease or uncontrolled diabetes mellitus
  15. Have a condition that the Investigator determines would significantly increase perioperative risk
  16. Any previous history of surgery on the posterior elements (laminectomy, posterior fusion) of the cervical spine
  17. Have metastatic malignant disease or active local malignant disease
  18. Have a life expectancy of less than 1 year
  19. Have an active systemic or local infection
  20. Have within 6 months of enrollment a significant untreated addiction to dependency producing medications or have been a substance abuser (including alcohol and illicit drugs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The intended study population is individuals who have been diagnosed with chronic, intractable pain of the upper limbs associated with a number of conditions, and who the Principal Investigator deems is an appropriate candidate for SCS therapy as required for this study.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2023-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Vallejo, MD, Study Chair — SGX Medical
Locations (1):
- SGX Medical, Bloomington, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1 subject was withdrawn by physician before starting the trial phase.
Pre-assignment Details: This is a single-arm observational study.
Groups:
- Subjects Treated With DTM SCS Programming: Subjects that met inclusion and exclusion criteria are trialed with DTM SCS programming.
Period: Prior to Trial Phase
Arm/Group | Subjects Treated With DTM SCS Programming
Started | 58
Completed | 57
Not Completed | 1
Not completed — Physician Decision | 1
Period: Trial Phase
Arm/Group | Subjects Treated With DTM SCS Programming
Started | 57
Completed | 52
Not Completed | 5
Period: Permanent Implant
Arm/Group | Subjects Treated With DTM SCS Programming
Started | 52
Completed | 46
Not Completed | 6
Period: 3 Months
Arm/Group | Subjects Treated With DTM SCS Programming
Started | 46
Completed | 43
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Subjects Treated With DTM SCS Programming
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 52
Upper Limb Pain [Mean (Standard Deviation); unit: units on a scale] — Visual Analog Score (0.0cm to 10.0cm). Higher score represents more pain.
  units on a scale | 7.25 (1.22)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Implanted Subjects Who Respond to DTM SCS Therapy at 3-months
Description: The primary efficacy endpoint is the percentage of implanted subjects who respond to DTM SCS therapy at 3-months after device activation. An individual responder is a subject that experiences at least a 50% decrease in upper limb pain relative to baseline assessment.
Time Frame: 3 months
Population: All subjects who receive a permanent SCS system implant. Does not include subjects that failed the trial phase nor subjects that did not receive permanent SCS system.
Measure: Number (95% Confidence Interval); unit: percentage of individual responder
Arm/Group | Subjects Treated With DTM SCS Programming
Number analyzed (Participants) | 43
percentage of individual responder | 100 [91.78 to 100]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Subjects Treated With DTM SCS Programming
All-Cause Mortality (participants affected / at risk) | 0/58
Serious Adverse Events (participants affected / at risk) | 1/58
Other Adverse Events (participants affected / at risk) | 3/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Treated With DTM SCS Programming (N=58)
Spinal cord bruising (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Treated With DTM SCS Programming (N=58)
Pocket Pain (Musculoskeletal and connective tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-30): https://cdn.clinicaltrials.gov/large-docs/11/NCT04466111/Prot_SAP_000.pdf